CLINICAL TRIAL: NCT06203275
Title: The G Protein-Coupled Receptor Kinase Type 2 Inhibitor Paroxetine as Adjunctive Therapy to Improve Insulin Sensitivity in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: aya ramadan ashmawy sarhan (Other)
Responsible Party: Sponsor-Investigator, aya ramadan ashmawy sarhan, tanta, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: paroxetine in type 2 diabetes
Record Dates: First submitted 2023-11-17; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GRK2 inhibitor; insulin resistance; diabetes; paroxetine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Diabetes Mellitus | interventions — Paroxetine

STUDY DESIGN:
Intervention Model Description: This proof of concept pilot study is designed as a randomized placebo controlled parallel trial. Forty four patients of both gender with confirmed diagnosis of T2DM will be randomized using sealed envelope method into two groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (control group) (Placebo Comparator): which will receive metformin based combined oral hypoglycemic plus placebo tablets
  Interventions: Drug: Placebo
- group II (intervention group) (Active Comparator): which will receive metformin based combined oral hypoglycemic plus 12.5 mg paroxetine daily at morning.
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Paroxetine — intervention group n=22 Patients with type 2 diabetes treated with metformin based combined oral hypoglycemic ( metformin plus DDP4 inhibitor or metformin plus sulfonylureas or metformin plus GLP-1 analogues) plus paroxetine 12.5 mg daily
  Arms: group II (intervention group)
Drug: Placebo — Patients with type 2 diabetes treated with metformin based combined oral hypoglycemic ( metformin plus DDP4 inhibitor or metformin plus sulfonylureas or metformin plus GLP-1 analogues) plus placebo daily
  Arms: group 1 (control group)

SUMMARY:
The aim of this study is to investigate the effect of GRK2 inhibitor paroxetine on insulin resistance in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (T2DM) is one of the most common metabolic disorders worldwide and its development is primarily caused by a combination of two main factors including defective insulin secretion by pancreatic β-cells and the inability of insulin sensitive tissues to respond to insulin.

Type 2 Diabetes Mellitus (T2DM) shares an intimate relationship with altered metabolism through the development of insulin resistance )IR(.

The G protein-coupled receptor kinase type 2 (GRK2) is involved in the regulation of many pivotal cell functions and is a key player in human health and diseases.In fact, GRK2 regulates insulin signaling through serine phosphorylated events. G protein-coupled receptor kinase type 2 up-regulation inhibits insulin signaling and glucose extraction due to a time dependent insulin-stimulated association of GRK2 with Insulin Receptor Substrate 1 (IRS1), leading to IRS1 serine phosphorylation and inactivation. Inhibition of hepatic GRK2 expression is sufficient to improve glucose homeostasis and insulin sensitivity, which eventually improves endothelial dysfunction in T2DM.

Preclinical studies reported that, genetic ablation of GRK2 in mice reduced insulin resistance. In this sense, inhibition of GRK2 activity could improve insulin sensitivity and might provide a new therapeutic target for the treatment of IR and T2DM. Paroxetine, an FDA-approved selective serotonin reuptake inhibitor (SSRI), was identified as a potent GRK2 inhibitor with higher selectivity for GRK2 over other GRKs both in vivo and in vitro.

Paroxetine binds to the active site of GRK2 and stabilizes the kinase domain in a conformation that inhibits G protein-coupled receptor (GPCR) phosphorylation and desensitization.6 A case report study demonstrated that during 3 months of paroxetine treatment, 35-year-old woman with poorly controlled T2DM experienced an increased frequency of hypoglycemic episodes. After discontinuation of paroxetine, her awareness of hypoglycemia was dramatically improved. The authors hypothesized that her hypoglycemic unawareness might be caused by autonomic dysfunction, which is an atypical manifestation of serotonin syndrome. Paroxetine also increased insulin sensitivity in non-diabetic patients who experienced remitted depression in a randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established diagnosis of type 2 diabetes.
* Patients with type 2 diabetes treated with metformin based combined oral hypoglycemic ( metformin plus DDP4 inhibitor or metformin plus sulfonylureas or metformin plus GLP-1 analogues)
* Glycated hemoglobin (HbA1c) ≥ 7% and ≤9
* Age between 20 and 65 years
* BMI ≥25 kg/m2

Exclusion Criteria:

* Pregnant and lactating women

  * Patients with diabetes complications except for hyperlipidemia if any.
  * Patients with acute or chronic illness (such as flu, cancer, rheumatoid arthritis, etc….)
  * Patients with renal impairment (S.Cr > 1.5 mg/dl) and hepatic impairment (Bilirubin level > 1.2 mg/dl).
  * Patients with cardiovascular diseases
  * Patients with condition that predispose to acidosis as COPD
  * Patients with glaucoma
  * Patients with thyroid disorders
  * Patients on the medications that affect carbohydrate metabolism such as beta blockers, contraceptives, thiazide diuretic, corticosteroids, sympathomimetic
  * Patients treated with any oral anti-diabetes agents other oral hypoglycemic agents or treated with insulin
  * Patients stabilized anticoagulants, antiplatelet, antipsychotics, MAOIs, amphetamines, NSAIDs, corticosteroids, ergotamine, levothyroxine, narcotic analgesic, tramadol, liver microsomal enzyme inhibitors and liver microsomal enzyme inducers

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the change in glycated Hemoglobin (HbA1c). | 3 months
Change in HOMA-IR . | 3 months

SECONDARY OUTCOMES:
The secondary outcome is the change in expression of GRK2 | 3 months